CLINICAL TRIAL: NCT02603263
Title: The Effect of a Descriptive Norm Promoting Vegetable Selection in a Workplace
Brief Title: The Effect of a Descriptive Norm Promoting Vegetable Selection in a Workplace Restaurant Setting: an Observational Study
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other); C H & Co Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UBirmingham-SNS7
Record Dates: First submitted 2015-10-22; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Eating Behaviour
Keywords: social norms; healthy eating; vegetables; field study
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Workplace Restaurant Customers: 1 Group (Workplace Restaurant Customers) across 3 sites (data to be combined at end of study)
  Study consists of three phases:
  1. Pre Intervention
  2. Intervention
  3. Post Intervention
  All phases lasted two weeks and included monitoring till receipts for meals (these were automatically generated and held on the tills electronically). The intervention phase consisted of posters being displayed in the restaurants, featuring a Social Norms Poster.
  Interventions: Other: Social Norms Poster

INTERVENTIONS:
Other: Social Norms Poster — A poster containing a social norms message: "Most people here choose to eat vegetables with their lunch"

SUMMARY:
Encouraging individuals to eat fruit and vegetables is difficult. However, recent evidence suggests that using social-based information might help. For instance, it has been shown that if people think that others are eating lots of fruit and vegetables, that they will consume more food to match the 'norm'.The purpose of this study was to determine whether social norm messages could be used to enhance vegetable purchases in workplace restaurants, in an observational study.

DETAILED DESCRIPTION:
In this study the investigators hypothesised that placing posters containing social norm messages promoting vegetable consumption in three workplace restaurants, would increase the purchase of meals with vegetables, and that this effect would be sustained over time. The investigators recruited three restaurants to this study. For two weeks (Pre-intervention phase) the investigators used till receipts to monitor the number of meals sold with or without vegetables at baseline. For the following two weeks (Intervention phase) the investigators placed social norms posters around the three restaurants, while continuing to collect till receipts. After this, the posters were removed, and receipts were monitored for a final two weeks (Post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Purchase of a meal at one of the restaurants

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Customers at workplace restaurants.
Sampling Method: Non-Probability Sample
Enrollment: 9445 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percentage of meals containing vegetables | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Thomas, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Thomas JM, Ursell A, Robinson EL, Aveyard P, Jebb SA, Herman CP, Higgs S. Using a descriptive social norm to increase vegetable selection in workplace restaurant settings. Health Psychol. 2017 Nov;36(11):1026-1033. doi: 10.1037/hea0000478. Epub 2017 May 25. PMID 28541071